CLINICAL TRIAL: NCT04774341
Title: Personalized Evidence-based Medicine Improves Outcomes of Anticoagulation Therapy in Patients With Atrial Fibrillation
Brief Title: Personalized Evidence-based Medicine in Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Center of Personalized Medicine, Pirogova (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other); I.M. Sechenov First Moscow State Medical University (Other); University of Rochester (Other); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Evgeny Pookushalov, Director for research and development, Center of Personalized Medicine, Pirogova
Other Study IDs: 20210225
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Adherence to Personalized EBM Anticoagulant Treatment in Patients at High Risk for Stroke
Keywords: Atrial fibrillation; Personalized evidence-based medicine; Clinical decision support systems; Stroke; Anticoagulation; Guidelines
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CDSS (MedicBK) Analysis
  Interventions: Drug: anticoagulation treatment
- Core Laboratory Analysis
  Interventions: Drug: anticoagulation treatment

INTERVENTIONS:
Drug: anticoagulation treatment — Adherence to personalized evidence-based anticoagulant treatment in patients at high risk for stroke with atrial fibrillation

SUMMARY:
A retrospective analysis

DETAILED DESCRIPTION:
4200 EMR of patients at high risk for stroke with 1-year follow-up will be enrolled in the current study and analyzed by clinical decision support systems (CDSS MedicBK) utilizing a core laboratory.

ELIGIBILITY:
Inclusion Criteria:

EMR only if an ECG diagnosis (12-lead ECG, 24-h Holter, or other electrocardiographic documentation) confirming AF was made in patients at high risk for stroke by CHA2DS2-VASc (≥2 in men and ≥3 in women).

Exclusion Criteria:

No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at high risk for stroke with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
The percentage of guideline-based and personalized EBM recommendations | 1-year
  The percentage of guideline-based and personalized EBM recommendations acted on by clinicians for anticoagulant therapy in patients with AF. All discrepancies between routine and CDSS-recommended treatment resulting in frame of guideline-based therapy and personalized EBM therapy will be adjudicated by core laboratory.

SECONDARY OUTCOMES:
Quantify the performance of the CDSS (MedicBK) algorithm | 1-year
  Quantify the performance of the CDSS (MedicBK) algorithm for presents treatment suggestions in frame of guideline-based therapy and personalized EBM therapy: the sensitivity, specificity, NPV, and PPV
1-year FU outcomes | 1-year
  Outcomes for all-cause mortality, thromboembolism (TE), bleeding, and the composite endpoint of any thromboembolism, cardiovascular death, or bleeding in relation to whether they were guideline-based treatment or personalized EBM treatment. Thromboembolism refers to stroke, transient ischemic attack, acute coronary syndrome, coronary intervention, cardiac arrest, peripheral embolism, and pulmonary embolism
Predictors | 1-year
  Predictors of guideline-based and personalized EBM adherence

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, Prof. MD PhD, Principal Investigator — Center for New Medical Technologies, Novosibirsk, Russia
Locations (1):
- Evgeny Pokushalov, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No